CLINICAL TRIAL: NCT00120679
Title: An Open-Label, Randomized Phase 2 Study to Validate a Patient Satisfaction Questionnaire for Anemia Treatment in Patient With Non-Small Cell Lung Cancer Treated With Darbepoetin Alfa or Recombinant Human Erythropoietin for Anemia Due to Chemotherapy
Brief Title: Treatment for Patients With Non-Small Cell Lung Cancer Who Developed Anemia Due to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020165
Record Dates: First submitted 2005-06-30; First posted 2005-07-19 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Non-Small Cell Lung Cancer; Anemia
Keywords: non-small cell lung cancer; darbepoetin alfa; Amgen
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa
Drug: recombinant human erythropoietin (rHuEPO)

SUMMARY:
The purpose of this study is to validate a Patient Satisfaction Questionnaire for Anemia Treatment (PSQ-AT) in non small cell lung cancer patients treated with darbepoetin alfa or recombinant human erythropoietin (rHuEPO) for anemia due to chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Subjects receiving multi-cycle chemotherapy for non-small cell lung cancer - Anemia due to chemotherapy (hgb less than or equal to 11.0 g/dL) - Expected to receive greater than or equal to 8 additional weeks of chemotherapy as part of their planned treatment - Karnofsky Performance Scale (KPS) greater than or equal to 50% - Adequate renal function - Adequate liver function Exclusion Criteria: - Iron deficiency - Unstable cardiac disease - Known positive test for human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2003-12

PRIMARY OUTCOMES:
Anemia correction

SECONDARY OUTCOMES:
Patient preference
Activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Schwartzberg LS, Yee LK, Senecal FM, Charu V, Tomita D, Wallace J, Rossi G. A randomized comparison of every-2-week darbepoetin alfa and weekly epoetin alfa for the treatment of chemotherapy-induced anemia in patients with breast, lung, or gynecologic cancer. Oncologist. 2004;9(6):696-707. doi: 10.1634/theoncologist.9-6-696. PMID 15561813
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com